CLINICAL TRIAL: NCT01127308
Title: An Open Label, Single-Period, Phase 1 Study To Evaluate The Pharmacokinetics, Excretion Balance And Metabolism Of [14C]-PF04971729 In Healthy Adult Male Subjects
Brief Title: A Radiolabeled Mass Balance Study of [14C]-Ertugliflozin (PF04971729, MK-8835) In Healthy Male Participants (MK-8835-038)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 8835-038
Record Dates: First submitted 2010-05-19; First posted 2010-05-20 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Absorption; Distribution; Metabolism; and Excretion; Mass Balance; Metabolic Profile; Radiolabel Study
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ertugliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [14C]Ertugliflozin (Experimental): Single dose - oral dosing suspension
  Interventions: Drug: Ertugliflozin

INTERVENTIONS:
Drug: Ertugliflozin — Ertugliflozin 25 mg will be administered as a single oral suspension containing approximately 100 uCi of [14C]ertugliflozin

SUMMARY:
This is single dose study of radiolabeled [14C]-ertugliflozin (PF04971729, MK-8835) in healthy male volunteers to study the absorption, distribution, metabolism and elimination of ertugliflozin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants with Body Mass Index of 17.5 to 30.5 kg/m2 and a total body weight >50 kg (110 lbs)

Exclusion Criteria:

* Female participants. Participants enrolled in a previous radionucleotide study or who have received radiotherapy or exposed to significant radiation within 12 months prior to screening

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2010-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Mean Percent of Dose Recovered in Urine and Feces Following a Single Oral Dose of [^14C]Ertugliflozin (100 µCi). | Up to 7 Days
Area under the plasma concentration-time curve (AUC) from time 0 to time of the last quantifiable concentration (AUClast) for ertugliflozin | Up to 7 Days
AUC from Hour 0 to infinity (AUCinf) for ertugliflozin | Up to 7 Days
Maximum plasma concentration (Cmax) of ertugliflozin | Up to 7 Days
Time taken to reach the maximum observed plasma concentration (Tmax) of ertugliflozin | Up to 7 Days
Ertugliflozin half life (t1/2) | Up to 7 Days
Amount of Ertugliflozin and metabolites in plasma, urine, and feces | Up to 7 Days
Number of Participants Experiencing an Adverse Event (AE) | Up to 7 Days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Fediuk DJ, Sahasrabudhe V, Dawra VK, Zhou S, Sweeney K. Population Pharmacokinetic Analyses of Ertugliflozin in Select Ethnic Populations. Clin Pharmacol Drug Dev. 2021 Nov;10(11):1297-1306. doi: 10.1002/cpdd.970. Epub 2021 Jul 2. PMID 34213819
- [Derived] Marshall JC, Liang Y, Sahasrabudhe V, Tensfeldt T, Fediuk DJ, Zhou S, Krishna R, Dawra VK, Wood LS, Sweeney K. Meta-Analysis of Noncompartmental Pharmacokinetic Parameters of Ertugliflozin to Evaluate Dose Proportionality and UGT1A9 Polymorphism Effect on Exposure. J Clin Pharmacol. 2021 Sep;61(9):1220-1231. doi: 10.1002/jcph.1866. Epub 2021 Jun 19. PMID 33813736